CLINICAL TRIAL: NCT02841813
Title: Genomic and Metabolomic Differences of Choline on the Risk of Preterm Delivery and Their Effects on Clinical Outcomes in Preterms Receiving Total Parenteral Nutrition Therapy
Brief Title: Effects of Genomic and Metabolomic Variations of Choline on Risk of Preterm Birth and Clinical Outcomes in Preterms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jie Zhu, Assitant Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-005
Record Dates: First submitted 2016-07-12; First posted 2016-07-22 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Genomic and Metabolomic Variations; Preterm Birth; Total Parenteral Nutrition
MeSH Terms: conditions — Premature Birth; Hyperphagia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples

GROUPS / COHORTS (4):
- The normal mothers group: No intervention
  Interventions: Other: No intervention
- The normal full-term infants group: No intervention
  Interventions: Other: No intervention
- The preterm mothers group: No intervention
  Interventions: Other: No intervention
- The preterms group: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The incidence of preterm birth increases annually. Premature delivery has become the leading cause of neonatal illness and death. For the survived premature babies, the incidence of sequelae is also higher than the full-term babies, which brings a heavy burden to a family and society. Preterm birth has become the important factor affecting the quality of births. The occurrence of premature birth is the outcome of combined action of genetic and environmental factors. However, its etiology is not clear. Recent studies have shown that the risk of preterm birth is associated with dietary factors. Choline is an essential nutrient for human health and it plays an important role in the growth and development of fetuses and neonates. The investigators previously found that serum levels of free choline in preterm mothers were lower than those in normal mothers with full-term birth. Serum levels of free choline also reduced in preterms after receiving parenteral nutrition (PN). However, the relationships between choline and preterm birth is not clear. Therefore, this study is aimed to explore the effect of choline intake during pregnancy and genetic polymorphisms on the risk of preterm birth and on the clinical outcomes in preterms receiving total PN therapy. Healthy Chinese pregnant women with their healthy term infants will be recruited as the control group, while Chinese women with preterm delivery and their preterm infants will be recruited as the preterm group. Dietary choline intake during pregnancy will be evaluated by semi-quantitative food frequency questionnaire and 24-h dietary recall questionnaire. Gene polymorphisms in the key enzymes of choline metabolism will be identified among the participated women and neonates through Real-time polymerase chain reaction. Choline and its related metabolites will be assayed using high performance liquid chromatography combined with mass spectrometry among all mothers and preterms before and after 7-days PN treatment. The influence of genetic risk factors and metabolic changes of choline on the physical and mental development of preterms will be evaluated. The results of this study will contribute to a comprehensive understanding of the role of choline and the relative gene polymorphisms on the risk of preterm birth, which will be helpful for estimating the high risk in advance. The results will also provide the scientific evidences to establish the personalized amount of choline intake among women and infants, optimize nutrition support for pregnant women and preterms, and promote better prenatal and postnatal care.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm group: preterm infants (gestational age < 37 w) and their mothers (125 pairs );
2. Control group: healthy full-term infants and their mothers (125 pairs );_
3. Admission to Xin Hua Hospital, Shanghai;_ 4.1600g ≤ birth weight ≤ 2100g for preterms;

5.Administration of total parenteral nutrition (TPN) ≥ 7d; 6.No contraindication of TPN therapy.

Exclusion Criteria:

1. Administration of TPN before enrollment;
2. Receive blood infusion during TPN treatment;
3. Liver or renal markers present at 2 times higher than the normal level;
4. Suspected or identified chromosome diseases, congenital metabolic disease, congenital digestive tract diseases and necrotizing enterocolitis;
5. Cytomegalovirus infection, viral hepatitis, and congenital or acquired immune deficiency.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy Chinese women with their healthy term infants were recruited as the control group, while Chinese women with preterm delivery and their preterm infants (gestational age < 37w) were recruited as the preterm group.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Distribution of single nucleotide polymorphisms of the targeted genes | June 2016 - December,2019
Plasma concentrations of choline | 3 years
Plasma concentrations of betaine | 3 years
Plasma concentrations of phosphocholine | 3 years

SECONDARY OUTCOMES:
Dietary questionnaire of choline intake during pregnancy | through study completion, an average of 3 years
Serum alanine aminotransferase | through study completion, an average of 3 years
Serum aspartate aminotransferase | through study completion, an average of 3 years
Serum total bilirubin | through study completion, an average of 3 years
Serum direct bilirubin | through study completion, an average of 3 years
Serum bile acid | through study completion, an average of 3 years
Serum gamma glutamyl transferase | through study completion, an average of 3 years
Serum triglyceride | through study completion, an average of 3 years
Mental developmental index | through study completion, an average of 3 years
Psychomotor developmental index | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhu, MD,PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China